CLINICAL TRIAL: NCT06746506
Title: Effect of Therapeutic Play With Amigurumi Toys During Blood Collection on Children's Pain and Fear
Brief Title: The Effect of Therapeutic Play Applied With Amigurumi Toys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Gamzegül ALTAY, Principal Investigator, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gamzegulaltay
Record Dates: First submitted 2024-12-17; First posted 2024-12-24 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Bloodletting
Keywords: bloodletting; fear; pain; children; amigurumi toy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amigurumi toy, pain and fear (Experimental)
  Interventions: Behavioral: Amigurumi toy
- control not pain and fear (No Intervention)

INTERVENTIONS:
Behavioral: Amigurumi toy — A toy prepared using anti-allergic yarn to suit children's developmental stages.
  Arms: Amigurumi toy, pain and fear

SUMMARY:
This study was planned to determine the effect of therapeutic play with amigurumi toys on pain and fear during blood collection in children aged 4 to 6 years who applied to the pediatric emergency department. The project is a randomized controlled trial. The study covers children aged 4-6 years who came to the blood collection unit of the pediatric emergency department of Recep Tayyip Erdoğan University Education and Research Hospital between January and June 2025. The research sample will consist of children who applied to the unit on the specified dates, met the research criteria, and volunteered to participate in the study. The "Survey Form", "Wong-Baker Facial Expression Assessment Scale" and "Child Fear Scale" will be used to collect data.

DETAILED DESCRIPTION:
Type of Study: The study is a randomized controlled trial. Population and Sample of the Research: The population of the research includes children aged 4-6 years who came to the pediatric blood collection unit of Recep Tayyip Erdogan University Training and Research Hospital pediatric emergency between January-June 2025.

The research sample; will consist of children who apply to the blood collection unit on the specified dates, meet the research criteria, and volunteer to participate in the study. The sample size of the study was calculated using the G*Power 3.1. 9.7 program. The results of the study titled "The Effect of Therapeutic Play Applied with Hand Puppets on Fear and Pain Due to Blood Collection in Preschool Children" by Oluç and Sarıalioğlu were used to determine the effect size of the study. In the calculation, the effect size was calculated as 0.71 (f = 0.71), 5% margin of error (α = 0.05) and 95% power (1-β = 0.95), and the sample size for each group was calculated as 40, and the study will be planned to be conducted with 80 children. It was decided to collect data from a total of 96 children (48 intervention, 48 control) by including a 20% spare sample in case of data loss.

In the study, "stratification and block randomization methods" will be used in assigning participants to control and intervention groups. It has been reported in the literature that variables such as age, gender and fear of interventional procedures are among the factors affecting the fear and anxiety experienced by children during interventional procedures. In this study, the variables of "age, gender and fear of blood collection" will be used in stratifying the children. Accordingly, the children will be stratified according to "age (4-5 and 6 years), gender (girls and boys) and fear of blood collection (fearful and not afraid)" and block randomization will be applied. In the study, 48 children will be included in each group by ensuring that the stratifications are repeated six times (2X3X2X4). The closed envelope method will be used to assign the stratified children to the control and intervention groups without bias. In the study, the data of each group will be collected on certain days of the week in order to prevent the child in one group from being affected by the procedure applied to the other group. The order of data collection of the groups will again be determined by the closed envelope method. The order of data collection for the control and intervention groups according to the days of the week will be as follows:

Toy group = Monday, Wednesday Control group = Tuesday, Thursday Data Collection Tools to be Used in the Research: Survey Form, Wong-Baker Facial Expression Assessment Scale and Child Fear Scale will be used to collect research data. Amigurumi toy will be used as an intervention tool in the research.

Survey Form: This form, prepared by the researcher by reviewing the literature, will include questions that include descriptive characteristics of the child.

Wong-Baker Facial Expression Assessment Scale (WB-YİDÖ): It was developed by Wong and Baker in 1981 and revised in 1983. This scale is used for pain diagnosis in children aged 3-18. This scale has six faces representing increasing pain intensity from zero to five from left to right. While the face on the far left has a smiling expression indicating a painless situation, the face on the far right has a crying expression corresponding to the most severe pain. The child is told to choose the face that best expresses his/her feelings. Six facial expressions are scored from left to right from 0 to 5 points (0 points = very happy/no pain, 5 points = most severe pain). As the score on the scale increases, pain tolerance decreases, and as the score decreases, tolerance increases.

Children's Fear Scale (CHS): The Child Fear Scale was developed by McMurty and colleagues in 2011 to measure fear in children undergoing painful medical procedures. The Child Fear Scale ranges from a neutral expression (0 = no anxiety at all) to a fearful face (4 = severe anxiety) Data Collection Before the researcher starts collecting data from the intervention and control group children, the children and their parents will be given preliminary information about the study (the purpose of the study, why the study is being conducted, the amigurumi toy will be used to relieve the child's pain and fear, etc.), and after obtaining verbal consent from the children and written consent from the parents, the data of the study will be obtained from the children who agree to participate in the study through face-to-face interviews. There are 4 nurses actively working in the blood collection department of the pediatric emergency unit where the study will be conducted. In order to eliminate differences in practice in this study, the blood collection procedures of all children participating in the study will be performed by the same nurse who has been working in the pediatric emergency department for 5 years. The parents of the children in all groups will be asked to accompany their children during the blood collection procedure. The children, their parents, and the nurse will be informed about the Wong-Baker Facial Expression Rating Scale and the Child Fear Scale.

Control Group: Before the blood collection procedure is performed in the control group, the pain and fear scales will be filled out by the nurse, child, and parent. Only routine practices will be performed. 5 minutes after the blood collection procedure, the pain and fear scales will be filled out again by the nurse, child and parent.

Intervention Group: Before the blood collection procedure, the pain and fear scales will be filled out by the nurse, child and parent. The child will be played with an amigurumi toy by the researcher during the procedure. 5 minutes after the blood collection procedure, the pain and fear scales will be filled out again by the nurse, child and parent.

Evaluation of Data The processing and statistical analysis of the collected data will be done with the analysis software called SPSS (Statistical Package for the Social Sciences) for Windows 20.0.

Ethical Principles of the Research In order to conduct the research, ethical approval (Number No: E-40465587-050.01.04-1230, Decision No: 2024/256) from the Ethics Committee of the Faculty of Medicine of Recep Tayyip Erdoğan University and official permission (Number No: E-64960800-799-251189932) from the relevant institution were obtained. The purpose of the study will be explained to the parents of the children who meet the research group criteria, the questions asked will be answered and their verbal and written consents will be obtained. Parents and children will be informed that the data collected during the research will be processed confidentially and anonymously, will not be used outside the study in question and that they can withdraw from the study at any time. Since the research is based on the use of data obtained from humans and therefore, due to the necessity of protecting personal rights, the relevant ethical principles of "Informed Consent", "Voluntariness" and "Protection of Confidentiality" will be followed. After the procedure is completed with the children in the control group, the "Equality Principle" will be tried to be fulfilled by playing with the toy.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6,
* Those who applied to the hospital as outpatients due to an acute illness,
* Those who were rated as yellow triage in the 3-level (red-yellow-green) triage system,
* Those whose mother or father was with the child during the procedure,
* Those whose blood was drawn with a single procedure,
* Those whose health status was stable will be included in the study.

Exclusion Criteria:

* - Children who have a history of sedative, analgesic or narcotic substance use within 24 hours before application,
* Children with a fever higher than 38 °C,
* Children with visual, hearing, language development, mental and neurological disorders,
* Children with a chronic or life-threatening disease,
* Children who refuse to participate in the study,
* Children who are treated in the red or green zone according to the triage system (red = critical emergency, requiring immediate action; yellow = unstable condition, requiring intervention within 60 minutes; and green = stable condition, intervention should be performed within 2 hours) will not be included in the study.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Wong-Baker Facial Expression Evaluation Scale | 6 months
  The scale was developed in 1981 and was revised in 1983. The scale is used to define pain in the 3-18 age group. The scale indicates that the severity of pain increases from zero to five as you go from left to right. Facial expressions are included under the numbers to describe the severity of pain. It consists of 6 faces in total. While the first smiling facial expression expresses the pain-free state, the crying facial expression at the end indicates the most severe pain intensity. While applying the scale, the child is told to choose the facial expression that best describes his feelings at the moment. Six facial expressions are scored between 0-5 points from left to right (0 points = very happy/no pain, 5 points = indicates the most severe pain). As the score obtained from the scale increases, the pain tolerance decreases, and as the score decreases, the tolerance increases.
Child Fear Scale | 6 months
  The scale was developed in 2011. The Child Fear Scale is used to determine the level of fear in children undergoing painful medical procedures. The Child Fear Scale is a scale from 0-4 showing five faces ranging from a neutral expression (0 = no worry) to the feared face (4 = serious anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, Güneysu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The aim is to share the research after it is published.